CLINICAL TRIAL: NCT04625764
Title: A Prospective, Open, Multi-center, Single-arm Study to Demonstrate the Feasibility of the CytoSorb® 300 mL Device to Remove Ticagrelor During Cardiopulmonary Bypass in Patients on Ticagrelor Undergoing Emergent Cardiothoracic Surgery
Brief Title: Ticagrelor Removal Study Using CytoSorb® 300 mL Device During CPB in Patients Undergoing Emergent Cardiothoracic Surgery
Acronym: CyTation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Corona pandemic, planned ammount of enrolled patient could not be reached, protocol section "Early termination of the study" - criterion "Difficulties in recruiting patients" is fully met->recruitment period will not be extended
Sponsor: CytoSorbents Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSI17
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Cardiopulmonary bypass; CPB; Ticagrelor removal; CytoSorb; Platelet reactivity; MEA platform test; Intensive care medicine; Hemadsorbtion; Extracorporeal blood purification; Coronary Artery Bypass Grafting; CABG; Cardiac Surgery; Aortic valve replacement; Mitral valve replacement
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients on ticagrelor undergoing emergent cardiothoracic surgery requiring CPB (Experimental)
  Interventions: Procedure: Blood sampling and analysis

INTERVENTIONS:
Procedure: Blood sampling and analysis — Blood sampling for pharmacokinetics (Plasma ticagrelor concentrations and its metabolite) and MEA platform testing (ADPtest, TRAPtest)

SUMMARY:
The aim of CyTation is to demonstrate intra-operative removal of ticagrelor by CytoSorb® hemadsorption in patients on ticagrelor undergoing emergent cardiothoracic surgery requiring CPB, using platelet reactivity to adenosine diphosphate (ADP) as a pharmacodynamics surrogate measure of ticagrelor levels in blood.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Males and females aged ≥18 years
* Patients treated with ticagrelor
* Emergency Coronary Artery Bypass Graft (CABG) surgery
* Cardiothoracic surgery requiring CPB ≤24 hours following the last dose of ticagrelor

Exclusion Criteria:

* Any cardiothoracic surgery >24 hours after last dose of ticagrelor
* Resuscitation
* Any pre-operative coagulopathy unrelated to ticagrelor or standard of care (SoC) to undergo surgery with CPB
* Sepsis (according to Sepsis 3.0 definition)
* Malignant tumor
* Left ventricular ejection fraction (LVEF) < 20%
* History or presence of significant pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, neurologic, or psychiatric disease which, in the opinion of the Investigator, increases risk to the patient or could confound the results of the study
* Presence of end-stage renal disease or currently receiving renal replacement therapy
* Patients with a history of major organ transplantation
* Patients in acute sickle cell crisis
* Patients concurrently requiring immunosuppressive therapy, with the exception of corticosteroids, or who are profoundly immune suppressed (e.g. CD4 < 200 or neutropenia with ANC < 1000/μL)
* Women of childbearing potential with a positive pregnancy test performed during the current admission or who are lactating. Women are considered not of child bearing potential if they have been sterilized at least 6 months prior to the study or if they are post-menopausal, defined as amenorrhea for at least 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity | 8 hours
  Proportion of patients with post-operative platelet reactivity to ADP above the level associated with increased bleeding risk (≥ 22 ADP-induced platelet aggregation units (AUC in units)) measured on the MEA platform immediately after CPB compared to immediately before CPB.

CONTACTS AND LOCATIONS:
Overall Officials: Kambiz Hassan, M.D., Principal Investigator — Asklepios Kliniken Hamburg gGmbH, Asklepios Klinik St. Georg, Abteilung für Herzchirurgie/ Chefarzt Prof. Michael Schmoeckel, Lohmühlenstr. 5, 20099 Hamburg/Germany
Locations (4):
- Germany (3):
  - University Hospital Essen, Essen
  - Asklepios Hospital St. Georg Hamburg, Hamburg
  - University Hospital Jena, Jena
- Institut National de Chirurgie Cardiaque et de Cardiologie Interventionnelle, Luxembourg, Luxembourg